CLINICAL TRIAL: NCT06957782
Title: The Value of 68Ga-FAPI PET/CT for Evaluating Peritoneal Treatment Response
Acronym: INTERACT-FAPI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, S. L. W. (Stijn) Koolen, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-520037-76-00
Record Dates: First submitted 2025-05-02; First posted 2025-05-05 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Peritoneal Metastasis; FAPI
Keywords: Peritoneal metastasis; Intraperitoneal; FAPI; PET/CT

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, single center, investigator-initiated, proof-of-concept, prospective imaging study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ⁶⁸Ga-FAPI-46 (Experimental): ⁶⁸Ga-FAPI-46 will be used as a diagnostic tracer for PET/CT to image peritoneal tumor cells.
  Interventions: Drug: ⁶⁸Ga-FAPI-46

INTERVENTIONS:
Drug: ⁶⁸Ga-FAPI-46 — All patients will be administered with 1.5 MBq/kg ⁶⁸Ga-FAPI-46. ⁶⁸Ga-FAPI-46 will be injected intravenously followed by a flush injection of 10 mL of saline following routine procedures.

SUMMARY:
Peritoneal metastases (PM), commonly originating from gastrointestinal and ovarian cancers, are associated with a poor prognosis and limited treatment options due to the diffuse nature of the disease and the inability of systemic chemotherapy to adequately penetrate the peritoneal surface. Intraperitoneal (IP) chemotherapy has emerged as a potential treatment modality for patients with extensive PM, allowing for higher local drug concentrations while minimizing systemic toxicity. However, current response evaluation methods, such as CT scans, have low sensitivity for detecting PM, and second-look laparoscopy, although more accurate, is invasive and unsuitable for repeated assessments. The ⁶⁸Ga-FAPI PET/CT scan offers a promising non-invasive alternative for assessing peritoneal response to IP chemotherapy. This imaging technique targets the fibroblast activation protein, which is overexpressed in cancer-associated fibroblasts within the tumor microenvironment. Early studies have shown that ⁶⁸Ga-FAPI PET/CT is a highly sensitive too in detecting peritoneal metastases. Given these advantages, the investigators hypothesize that ⁶⁸Ga-FAPI PET/CT could improve the evaluation of treatment response in patients undergoing IP chemotherapy for PM, offering a non-invasive and accurate alternative to current methods. The primary objective of this study is to investigate the accuracy of ⁶⁸Ga-FAPI PET/CT for evaluating peritoneal response in patients with peritoneal metastases undergoing repeated IP chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* A planned start of repeated IP chemotherapy (with or without the combination of systemic chemotherapy) for macroscopic peritoneal metastases;
* WHO-performance score of 0 to 1;
* Aged 18 years or older;
* Written informed consent according to the ICH-GCP and national/local regulations.

Exclusion Criteria:

* Impaired renal function, defined as eGFR <25 ml/min/1,73 m2. An exception can be made in consultation with the treating physician;
* Pregnancy/breastfeeding. For the latter, temporary discontinuation may be considered;
* Known allergic reaction to therapeutic radiopharmaceuticals;
* Inability to lie still on the back for the duration of PET-CT;
* Any (other) condition, disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that may affect the interpretation of the results, or which might contribute substantially to the patient's experience of study burden (such as non-suppressible claustrophobia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy of ⁶⁸Ga-FAPI | 18 weeks
  To investigate the accuracy of the ⁶⁸Ga-FAPI PET/CT for peritoneal response evaluation in patients with peritoneal metastases that are treated with any form of repeated IP chemotherapy. The accuracy will be calculated as the sensitivity and specificity of the ⁶⁸Ga-FAPI PET/CT with clinical assessment during MTB and/or histopathological outcome at second laparoscopy as a reference standard.

SECONDARY OUTCOMES:
Tumor response to IP chemotherapy | 18 weeks
  To measure the tumor response to IP chemotherapy. The absolute change in peritoneal tumor size or volume as measured by imaging before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Koolen, PharmD, PhD, Principal Investigator — Erasmus Medical Center

IPD SHARING:
Plan to Share IPD: No